CLINICAL TRIAL: NCT01845584
Title: NPB-01(Intravenous Immunoglobulin) Therapy for Patients With Anti-aquaporin 4 Antibody Positive Neuromyelitis Optica Spectrum Disorder Not Provided Adequate Effect of Therapy to Steroids Plus Therapy.
Brief Title: Phase II Clinical Trial of NPB-01 in Patients With Anti-aquaporin 4 Antibody Positive Neuromyelitis Optica Spectrum Disorder Not Provided Adequate Effect of Therapy to Steroids Plus Therapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPB-01-08/E-01
Record Dates: First submitted 2013-04-26; First posted 2013-05-03 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: IVIG in Neuromyelitis Optica spectrum disorder; Patients with Neuromyelitis Optica spectrum disorder
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPB-01 (Experimental): Intravenous immunoglobulin
  Interventions: Drug: NPB-01

INTERVENTIONS:
Drug: NPB-01
  Other Names: Intravenous immunoglobulin

SUMMARY:
Patients diagnosed with anti-aquaporin 4 antibody positive Neuromyelitis Optica spectrum disorder were confirmed based on diagnostic criteria. Patients who meet all inclusion criteria and do not conflict with the exclusion criteria will receive steroid plus therapy （1g/day for five consecutive days）. Subsequently, patients who not provided adequate effect of therapy to steroids plus therapy will receive NPB-01 (intravenous immunoglobulin) 400mg/kg/day for five consecutive days. Patients evaluated Quantification of nerve and spinal cord impairment （QOSI） and the Expanded Disability Status Scale （EDSS）/ Functional Systems （FS） and anti-aquaporin 4 antibody et al.

As a safety endpoint, the safety of NPB-01 will be investigated the occurrence of adverse events by one year after the start of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who become positive for anti-aquaporin 4 antibody or have becomed.
2. Patients who have developed myelitis.
3. Patients who run beyond greater than 30 days at least from last time in relapse.
4. Patients who new neurological symptom or worsening neurological symptom or flared neurological symptom have sustained 24 hours at least not associated fever or infection.
5. Patients who have an acute exacerbation at informed consent.
6. Patients who need steroid plus therapy（1g/day for five consecutive days）.
7. Patients who can start steroid plus therapy within 3 days after informed consent.
8. Patients who be inadequate to effect to steroid plus therapy.
9. Patients with greater than or equal to twenty years old at informed consent.

Exclusion Criteria:

1. Patients who have developed optic neuritis.
2. Patients treated with intravenous immunoglobulin within 14 days before informed consent.
3. Patients with malignancy at informed consent.
4. Patients with history of shock or hypersensitivity for NPB-01.
5. Patients with IgA deficiency.
6. Patients with impaired liver function.
7. Patients with impaired renal function.
8. Patients with cerebro- or cardiovascular disorders.
9. Patients with high risk of thromboembolism.
10. Patients with hemolytic/hemorrhagic anemia.
11. Patients with decreased cardiac function.
12. Patients with decreased platelet.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Quantification of nerve and spinal cord impairment （QOSI） at 29 days | 29 days
Change from Baseline Expanded Disability Status Scale （EDSS）/ Functional Systems （FS） at 29 days | 29 days
Change from Baseline anti-aquaporin 4 antibody at 29 days | 29 days

CONTACTS AND LOCATIONS:
Locations (1):
- Japan, Osaka, Japan